CLINICAL TRIAL: NCT06693830
Title: Sequencing-guided cHemotherapy Optimization Using Real-Time Evaluation in Newly Diagnosed DLBCL With Circulating Tumor DNA: SHORTEN-ctDNA
Brief Title: ctDNA-guided Therapy Optimization in Newly Diagnosed DLBCL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hua-Jay J Cherng, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Conquer Cancer Foundation (Other); Foresight Diagnostics (Unknown)
Responsible Party: Sponsor-Investigator, Hua-Jay J Cherng, MD, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: AAAU9823; R03CA286676 (NIH)
Record Dates: First submitted 2024-11-15; First posted 2024-11-18 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; Lymphoma, B-Cell; Diffuse Large B Cell Lymphoma; Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; High-grade B-cell Lymphoma
Keywords: circulating tumor DNA; measurable residual disease
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Neoplasm, Residual

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Group 1 (Other): All participants on this study will receive standard immunochemotherapy treatment for the first 4 cycles. Blood samples will be collected for real-time ctDNA sequencing with the PhasED-seq assay.
  Participants with undetectable ctDNA from the first day of cycle 4 and in a complete response (CR) on their PET/CT scan will get de-escalated treatment for cycle 5 and cycle 6 (rituximab alone without chemotherapy)
  Interventions: Device: Phased Variant Enrichment and Detection Sequencing (PhasED-seq); Other: De-escalated Treatment
- Group 2 (Other): All participants on this study will receive standard immunochemotherapy treatment for the first 4 cycles. Blood samples will be collected for real-time ctDNA sequencing with the PhasED-seq assay. Participants with detectable ctDNA, not in in a CR on PET/CT, and/or whose ctDNA sequencing was unsuccessful for any reason will continue standard of care for the remainder of treatment (cycle 5 and 6).
  Interventions: Device: Phased Variant Enrichment and Detection Sequencing (PhasED-seq); Other: Standard of Care Treatment

INTERVENTIONS:
Device: Phased Variant Enrichment and Detection Sequencing (PhasED-seq) — PhasED-seq designed to detect minimal residual disease (MRD) as indicated by the presence of circulating tumor DNA (ctDNA) evidenced by an aggregate signal of phased variants (PVs) in the plasma of patients diagnosed with large B-cell lymphoma (LBCL) following first-line therapy.
Other: Standard of Care Treatment — Standard of Care Treatment for cycles 1-6
  Arms: Group 2
Other: De-escalated Treatment — Standard of Care Treatment for cycles 1-4 and de-escalated treatment for cycles 5 and 6
  Arms: Group 1

SUMMARY:
The purpose of this study is to 1) determine whether it is feasible to measure circulating tumor DNA (ctDNA) in real-time during standard treatment for newly diagnosed diffuse large B-cell lymphoma (DLBCL), and 2) evaluate the outcomes of participants with undetectable ctDNA in the middle of treatment who receive a shortened course of chemotherapy.

There are no investigational drug agents to be administered in this study. The investigational assay, phased variant enrichment and detection sequencing (PhasED-seq) will be used to guide de-escalation of standard-of-care therapy for newly diagnosed DLBCL.

The PhasED-seq assay has not yet been approved by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
The feasibility of real-time ctDNA sequencing with PhasED-seq during DLBCL therapy has yet to be established. There are logistical challenges to developing a consistent and efficient workflow for obtaining, processing, and sequencing patient samples during frontline immunochemotherapy. ctDNA sequencing must be reliable with a low failure rate before it can be adopted as an integral biomarker for treatment decision making in the clinic. Furthermore, the outcomes of patients who have undetectable ctDNA with PhasED-seq during treatment who de-escalate their chemotherapy must be assessed.

In this study an anticipated 40 patients with newly diagnosed DLBCL will be screened for a target enrollment goal of 32 participants. These 32 patients will receive standard treatment with 4 cycles of R-CHOP or R-pola-CHP immunochemotherapy. These patients will have blood samples collected after 3 cycles to test for the presence of ctDNA in real-time. Patients who have successful real-time sequencing and have undetected ctDNA as well as a complete remission on interim re-staging scans will de-escalate treatment and omit chemotherapy for their final 2 cycles of treatment. These patients will receive rituximab alone for their final 2 cycles. All others will continue standard treatment.

26 participants are expected to have successful real-time sequencing, of which 13 patients are expected to meet criteria for treatment de-escalation and omit chemotherapy for their final 2 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed, histologically confirmed CD20+ DLBCL

   * Stage II-IV disease
   * Planned for anthracycline-based therapy with standard dosed R-CHOP or R-pola- CHP without consolidative radiation
   * Measurable disease on cross sectional imaging ≥ 1.5 cm in longest diameter and measurable in two perpendicular dimensions, with at least one corresponding hypermetabolic lesion by Lugano classification on baseline FDG PET/CT or CT with intravenous contrast of the chest, abdomen, and pelvis if FDG PET/CT not available.
2. Age 18 years or older at time of screening
3. Subject/legal representative willing and able to provide written informed consent
4. Ability to comply with outpatient treatment, laboratory monitoring, and required clinic visits for duration of study participation
5. Organ function as assessed by laboratory and cardiac function testing and Eastern Cooperative Oncology Group (ECOG) performance status in appropriate range for receipt of R-CHOP or R-pola-CHP at standard dose as per treating physician

Exclusion Criteria:

1. Previous treatment for diffuse large B-cell lymphoma, except as outlined below:

   * Up to 14 days of corticosteroids for the relief of lymphoma-related symptoms
   * A dose of pre-phase vincristine or rituximab
   * One cycle of R-chemotherapy (including but not limited to R-CHOP, R-pola-CHP, dose-adjusted etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin, rituximab [DA-EPOCH-R) that has not started more than 28 days prior to consent
   * Intrathecal chemotherapy for central nervous system (CNS) prophylaxis
   * Radiation therapy for the treatment or prevention of spinal cord compression that has not started more than 28 days prior to enrollment
2. Simultaneous participation in other treatment clinical protocol
3. Planned anti-lymphoma therapies beyond R-CHOP or R-pola-CHP:

   * Consolidative radiation to any baseline sites of disease
   * Planned high-dose intravenous methotrexate for central nervous system (CNS) lymphoma prophylaxis (both mid-cycle and EOT excluded)

     * Any number of doses of intrathecal chemotherapy for CNS lymphoma prophylaxis are allowed
4. Transformed indolent lymphoma (including follicular lymphoma, marginal zone lymphoma, or lymphoplasmacytic lymphoma) or grade IIIB follicular lymphoma
5. Known CNS involvement by lymphoma. R-CHOP and R-pola- CHP are insufficient to treat CNS disease.
6. Any disease characteristics that would make R-CHOP or R-pola-CHP without radiation insufficient therapy at the discretion of the treating physician

   * High-grade B-cell lymphoma with rearrangement of MYC and BCL2, primary mediastinal B-cell lymphoma, and HIV-associated lymphomas are excluded
7. Richter transformation of chronic lymphocytic leukemia
8. Pregnancy and/or nursing period. R-CHOP and R-pola-CHP may cause fetal harm or birth defects, and effects of exposure in the breastfed infant are unknown.

   * A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "childbearing potential"
   * Women of childbearing potential are eligible if a negative serum or urine beta human chorionic gonadotropin pregnancy test is documented within 28 days of screening, and they must agree to us an effective contraception method during systemic treatment
   * Men who have partners of childbearing potential must agree to use an effective contraceptive method during systemic treatment
   * In addition to routine contraceptive methods, "acceptable contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen.
9. Uncontrolled active systemic infection

   * Patients with a positive hepatitis B virus (HBV) core antibody and negative HBV surface antigen consistent with prior HBV exposure must be willing to take appropriate anti-viral prophylaxis.
   * Patients with evidence of chronic HBV infection must have undetectable HBV viral load on the most recent test results obtained within the last year and received suppressive therapy.
   * Participants with a history of hepatitis C virus (HCV) infection must have an undetectable viral load. Participants currently being treated for HCV infection must have undetectable HCV viral load test on the most recent test results obtained within 28 days prior to consent.
10. Active second malignancy unless in remission and with life expectancy > 2 years with exception of patients diagnosed with basal cell or squamous cell carcinoma of the skin or carcinoma "in situ" of the cervix or breast who are eligible even if diagnosed within 2 years. If patients have another malignancy that was treated within the last 2 years, such patients may be enrolled, if the likelihood of requiring systemic therapy for this other malignancy within 2 years is less than 10%, as determined by an expert in that particular malignancy at CUIMC, and after consultation with the Principal Investigator. Hormone therapy for treated prostate and breast cancer is allowed.
11. Known hypersensitivity to any component of R-CHOP or R-pola-CHP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Success Rate of Real-Time Circulating Tumor DNA (ctDNA) Sequencing | up to 5 months
  Success defined as: C4D1 sample collected, DNA successfully sequenced from the diagnostic tissue sample, C4D1 timepoint result must be available within 28 days of C4D1
Complete Response Rate (CRR) | up to 6 months
  Complete response rate as assessed by PET/CT scan in participants who receive de-escalated treatment

SECONDARY OUTCOMES:
Rate of Minimal Residual Disease (MRD) Negativity | Up to 4 months
  MRD negativity defined as ctDNA negativity as determined by blood sample analysis
Time to ctDNA Result | Up to 28 days
  Time from sample collection to ctDNA result
Proportion of Participants Eligible for De-escalation | Up to 5 months
  The proportion of participants eligible for de-escalation
Progression Free Survival (PFS) Rate | 2 years
  PFS defined as the time between C1D1 of therapy and progression of DLBCL.
Overall Survival (OS) Rate | 2 years
  OS defined as the time between C1D1 of therapy and death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Hua-Jay J Cherng, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States